CLINICAL TRIAL: NCT05529615
Title: Circulating Tumor DNA Guided Adjuvant Chemotherapy for Colon Cancer: A Prospective, Multicenter, Open-label, Randomized Controlled Clinical Trial
Brief Title: Circulating Tumor DNA Guided Adjuvant Chemotherapy for Colon Cancer
Acronym: CTAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Aiwen Wu, Director of GI cancer III, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PKUCH-C03
Record Dates: First submitted 2022-08-25; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Colon Cancer; Circulating Tumor DNA
Keywords: chemotherapy; ctDNA; colon cancer; prognosis
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stage II with high risk and stage III with low risk（T1-3N1） (Other): ctDNA will be detected at 7 days after surgical treatment. If，ctDNA(-)-> observation； ctDNA(+)-> 1:1 randomized as Capeox chemotherapy 3 months and observation. CtDNA will be detected at 4 months after surgical treatment.
  Interventions: Procedure: detection of ctDNA
- stage III with high risk（T4 or N2 or both） (Other): ctDNA will be detected at 7 days after surgical treatment. All the stage III with high risk will receive Capeox chemotherapy 3 months. ctDNA will be detected after the completion of Capeox chemotherapy 3 months. If，ctDNA(-) -> observation； ctDNA(+) -> 1:2 randomized as Capeox chemotherapy 3 monthsand second line treatment（decided by physician）.
  CtDNA will be detected at 7 months after surgical treatment.
  Interventions: Procedure: detection of ctDNA

INTERVENTIONS:
Procedure: detection of ctDNA — the ctDNA will be detected during the treatment and served as the andomization basis

SUMMARY:
The IDEA study classified stage III colon cancer into low-risk (T1-3/N1) and high-risk patients (T4 or N2) according to TNM stage. The results showed that for some low-risk patients, chemotherapy could be reduced without survival loss.

In recent years, circulating tumor DNA had achieved encouraging results in monitoring recurrence and metastasis after surgery, and has potential clinical application value. Postoperative ctDNA is also considered as a marker of increased risk of recurrence for stage I-III colon cancer and can provide predictive information for decision making on adjuvant treatment.

The results of GERCOR-PRODIGE, concomitant study of IDEA-FRANCE, showed that in the high-risk group, the patients with ctDNA positive and receiving adjuvant chemotherapy for 6 months had similar prognosis as the patients with ctDNA negative and receiving chemotherapy for 3 months; in the low-risk group, the patients with ctDNA positive but receiving chemotherapy for 3 months had worst prognosis, and the prognosis of patients with ctDNA negative chemotherapy for 3 months and 6 months and ctDNA positive chemotherapy for 6 months were similar. This indicates that risk stratification can be further performed according to the results of ctDNA after clinical pathological staging. Pathological staging is still an important decision-making factor for chemotherapy. It is not reliable to the chemotherapy decision making just based on ctDNA and abandoning clinical staging.

Therefore, a prospective, multicenter, open-label, randomized controlled clinical trial was designed aimed to investigate circulating tumor DNA guided adjuvant chemotherapy for colon cancer. In this study, all the patients are divided into high-risk group and low-risk group according to the postoperative pathology. Patients in each group were randomized to different treatment schedule according to the results of ctDNA.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75
2. Colon adenocarcinoma confirmed by pathology (including high and high differentiated tubular adenocarcinoma, papillary adenocarcinoma, low differentiated adenocarcinoma, mucinous adenocarcinoma and signet ring cell carcinoma)
3. Postoperative pathology is stage II with high-risk factors or stage III;

   High risk stage II refers to stage II colon cancer with at least one of the following:

   a) T4 stage; b) The number of lymph nodes detected was less than 12; c) Poor differentiation (except MSI-H); d) Complicated with LVI or PNI；e) Complicated with obstruction or perforation.
4. No distant metastasis was found in preoperative imaging examination and operation;
5. ECOG score: 0-2 points;
6. MSS/pMMR and BRAF wild type
7. Start time of chemotherapy is less than 2 months from the operation
8. Have sufficient organ functions;
9. The baseline blood routine and biochemical indexes of the subject meet the following standards:

   * hemoglobin ≥ 9.0 g / dl;
   * absolute neutrophil count (ANC) ≥ 1500 / mm3;
   * platelet count ≥ 100000 / mm3;
   * total bilirubin ≤ 1.5 times the upper limit of normal value (ULN);
   * glutamic pyruvic transaminase and glutamic oxalic transaminase ≤ 2.5 times ULN;
   * creatinine ≤ 1.5 times ULN;
10. Patients or family members who can understand the study protocol and are willing to participate in the study shall provide written informed consent.

Exclusion Criteria:

1. Receive chemotherapy, radiotherapy or immunotherapy before operation
2. History of malignant tumor in the past 5 years (except fully cured cervical carcinoma in situ or basal cell carcinoma or squamous epithelial cell skin cancer)
3. Pregnant women
4. Serious mental illness
5. Those with poor physical condition and difficult to complete chemotherapy
6. Patients or family members cannot understand the conditions and objectives of this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2684 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival rate | 3 year
  Whether the 3-year DFS of ctDNA negative colon cancer patients in the low-risk group is not inferior to adjuvant chemotherapy; 2) Whether second-line chemotherapy can significantly improve the 3-year DFS of ctDNA positive colon cancer patients in the high-risk group compared with standard chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Aiwen Wu, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking university cancer hospital, Beijing, Beijing Municipality, China